CLINICAL TRIAL: NCT04253314
Title: Prospective Multi-Center Observational Study to Assess Effectiveness of Venclexta (Venetoclax) in Acute Myeloid Leukemia (AML) Patients Ineligible for Standard Induction Therapy in Routine Clinical Practice in Russian Federation (INNOVATE)
Brief Title: A Study of the Effectiveness of Venetoclax Tablets in Adult Acute Myeloid Leukemia Participants Ineligible for Standard Induction Therapy in Russian Federation
Acronym: INNOVATE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-147
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Acute Myeloid Leukemia (AML); Venetoclax; Venclexta
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Venetoclax Participants: Participants treated with Venetoclax in accordance with approved local label. Decision to treat with Venetoclax was made prior to offering participation in this study.

SUMMARY:
Acute Myeloid Leukemia (AML) is a cancer of the blood and bone marrow and is the most common acute leukemia in adults. This study will evaluate how well Venetoclax works to treat AML in adult participants who are ineligible for standard induction therapy in Russian Federation.

Venetoclax is a drug approved to treat Acute Myeloid Leukemia. All study participants will receive Venetoclax as prescribed by their study doctor in accordance with approved local label. Adult participants with a diagnosis of AML who are ineligible for standard induction therapy will be enrolled. Around 50 participants will be enrolled in the study in approximately 15 sites in Russian Federation.

Participants will receive venetoclax tablets to be taken by mouth daily according to the approved local label. The duration of the study is approximately 18 months.

There is expected to be no additional burden for participants in this trial. All study visits will occur during routine clinical practice (approximately every 3 months) and participants will be followed for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed acute myeloid leukemia (AML) (de novo or secondary) and eligible to receive Venetoclax as per Russian Ministry of Health label
* Ineligible for standard induction therapy with cytarabine and anthracycline
* Eastern Cooperative Oncology Group (ECOG) score >2
* White blood cell counts <25 x 109 per liter
* Started Venetoclax within 4 weeks of enrolling in study

Exclusion Criteria:

* Acute promyelocytic leukemia
* Contraindications to Venetoclax as listed on the approved local label in Russian Federation
* Neuroleukemia - active central nervous system (CNS) involvement
* Participation in a clinical trial with an investigational drug for AML within 30 days prior to Venetoclax treatment initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with acute myeloid leukemia (AML) treated with Venetoclax per approved local label in Russian Federation.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Approximately 18 months
  Defined as the time (in days) between the date of first Venetoclax intake to date of death.

SECONDARY OUTCOMES:
Overall Response Rate | Approximately 18 months
  Defined as the percentage of participants with either complete response (CR) or complete response with incomplete hematological recovery (CRi) according to physician's assessment.
Best Overall Response Rate | Approximately 18 months
  Defined as the percentage of participants with either CR or CRi according to physician's assessment during Venetoclax treatment.
Best complete Remission | Approximately 18 months
  Defined as the percentage of participants with CR according to physician's assessment during Venetoclax treatment.
Time to First Response | Approximately 18 months
  Defined as the time (in weeks) between the date of first Venetoclax intake to first response, among CR, CRi, and morphologic leukemia free state (MLSF).
Time to Best Response to Treatment | Approximately 18 months
  Defined as the time (in weeks) between the date of first Venetoclax intake and the date of hte assessment having documented the best response among CR, CRi, and MLSF.
Duration of Response (DOR) | Approximately 18 months
  Defined as the time (in weeks) between the date of the first assessment documenting the response to Venetoclax (either CR, CRi, or MLSF) and the date of the first assessment having documented the progression.
Event-Free Survival (EFS) | Approximately 18 months
  Defined as the time (in weeks) between the date of first Venetoclax intake and the date of the first assessment having documented disease progression (primary refractory disease, or relapse from CR, CRi, or death from any cause).
Relapse-Free Survival (RFS) | Approximately 18 months
  Defined as the time between the date of CR and the date of the first assessment having documented disease progression or death from any cause.
Time to Transfusion Independence | Approximately 18 months
  Defined as the time (in weeks) between the date of first Venetoclax intake and the absence of any red blood cell (RBC) or platelet transfusion during any consecutive 8 weeks during the treatment period.
Percentage of participants treated with Venetoclax in combination with hypomethylating agents (HMAs) | Approximately 18 months
  Defined as the percentage of participants treated with Venetoclax in combination with hypomethylating agents (HMAs).
Percentage of participants treated with Venetoclax in combination with low dose cytarabine (LDAC) | Approximately 18 months
  Defined as the percentage of participants treated with Venetoclax in combination with low dose cytarabine (LDAC).
Percentage of participants treated with Venetoclax in combination with other therapeutic agents | Approximately 18 months
  Defined as the percentage of participants treated with Venetoclax in combination with other therapeutic agents
Percentage of participants with dose modifications | Approximately 18 months
  Percentage of participants with dose modifications.
Percentage of participants with dose interruptions | Approximately 18 months
  Percentage of participants with dose interruptions
Percentage of participants taking concimtant CYP3A medications | Approximately 18 months
  Percentage of participants taking concimtant CYP3A medications while treated with Venetoclax.
Number of participants with adverse events | Approximately 18 months
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity after the first dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- Russia (10):
  - Moscow State budget healthcare /ID# 218569, Moscow, Moscow
  - Saratov State Medical University n.a. V.I. Razumovskiy /ID# 226059, Saratov, Saratov Oblast
  - Hematology department State budgetary health care institution Volgograd region /ID# 229813, Volgograd, Volgograd Oblast
  - Regional Clinical Hospital of Irkutsk /ID# 218570, Irkutsk
  - Clinical Medico-Sanitary Unit #1 /ID# 222502, Perm
  - Russian Research Institute of Hematology and Transfusiology of the FMBA /ID# 229812, Saint Petersburg
  - R.M.Gorbacheva Research Institute of Paediatric Oncology, Haematology and Transp /ID# 224831, Saint Petersburg
  - Almazov National Medical Research Centre /ID# 218571, Saint Petersburg
  - Republican Hospital #1 - National Center of Medicine of Sakha (Yakutia) /ID# 224830, Yakutsk
  - Sakhalin Regional Clinical Hospital /ID# 222501, Yuzhno-Sakhalinsk

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P20-147#additional-resources-section